CLINICAL TRIAL: NCT00526266
Title: Evaluating Physiological Markers of Emotional Trauma: A Randomized Controlled Comparison of Mind-Body Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Principal Investigator, Dawson Church, Executive Director, Soul Medicine Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ROM-ACEP-SMI-IMCSR-1
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Hypermobility, Joint; Depression; Anxiety
MeSH Terms: conditions — Joint Instability; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Emotional Freedom Techniques (EFT)
- 2 (Placebo Comparator)
  Interventions: Behavioral: Diaphragmatic Breathing (DB)
- 3 (No Intervention): No Treatment

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques (EFT) — A half hour treatment with EFT following a standardized protocol. Both Range of Motion (ROM) physical issues are treated with EFT, as well as any possible emotional issues underlying limited ROM.
  Arms: 1
Behavioral: Diaphragmatic Breathing (DB) — Diaphragmatic Breathing (DB) instead of EFT tapping, but with all the "Setup Statements" and components of the Experimental Group, with the exception of tapping. DB is substituted for tapping.
  Arms: 2

SUMMARY:
The purpose of the study is to determine if a physiological marker, joint rotation of the upper body, can be affected by the release of emotional trauma during a brief psychotherapeutic encounter, and whether acupressure is an active ingredient in EFT.

DETAILED DESCRIPTION:
The effect of emotional trauma on physiological functioning has been documented in a number of studies. The largest of these is the ACE study, (ACE=Adverse Childhood Experiences), which examined the health outcomes of over 17,000 patients at Kaiser Permanente Hospitals. It was performed by Kaiser in collaboration with the Centers for Disease Control, on a population with a median age of 56. The ACE study found that those patients with a high incidence of Adverse Childhood Experiences or ACEs had higher rates of bone fractures, cancer, heart disease, hypertension, depression, smoking, suicide, diabetes, and other physical and psychological ailments. The authors of the study compared the health care system's focus on treating disease in adults to a fire brigade directing their water at the smoke, rather than at the originating fire. They recommended that health care providers focus on the emotional trauma which they believe contributes to many illnesses.

The current study seeks to determine if the treatment of emotional trauma has an effect on physiological function. As a marker of physiological function, the authors of this study have chosen the range of motion of the joints of the upper body. Shoulder joint stiffness and syndromes such as frozen shoulder typically take months or even years to heal, and rapid resolution is unusual, though most such injuries do indeed heal over time. Range of motion is a convenient marker of physiological change because it can be measured accurately in degrees using a goniometer, a protractor-like device routinely used in occupational therapy and physical therapy. Changes after treatment can be immediately noted.

The emotional trauma treatment modalities being investigated are Emotional Freedom Techniques or EFT, and Diaphragmatic Breathing or DB, with the DB group receiving an identical protocol but with DB substituted for the acupressure component of EFT. They are being compared with a no treatment control group. Studies of EFT have shown this therapy to be effective in removing or reducing emotional traumas, such as phobias, in a single brief treatment session, as well as in reducing anxiety. The effects hold over time. Most prior studies using EFT as a treatment modality study the effects of only one session, and have found that EFT can be effective even with a very brief course of treatment. For the current study, one 30 minute EFT treatment is undertaken. The range of motion of the shoulder joint is recorded before and after treatment by a licensed occupational therapist using a goniometer. The Diaphragmatic Breathing protocol used by the second group has a verbal content identical to the EFT group, but substitutes DB for acupressure. A follow up assessment of subjects is done after 30 days. Range of motion usually does not relapse, but instead becomes greater, following conventional treatments, and this measure has the advantage of requiring a relatively short follow up period, rather than the longer period required for other physiological markers.

The purpose of the study is to discover if a significant change in the range of motion occurs after treatment, and to dismantle the acupressure from the verbal component of EFT by substituting DB for this portion of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Limited Range of Motion (ROM) of a joint in the upper body

Exclusion Criteria:

* Post-operative recovery
* Receiving rehabilitation treatment
* Under psychiatric care
* Currently using prescription psychotropic medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-09; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Mental Health Symptoms | One Treatment Session

SECONDARY OUTCOMES:
Range of Motion (ROM) of joints of the upper body | Before and immediately after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Principal Investigator — Soul Medicine Institute
Locations (1):
- Integrative Medical Clinic of Santa Rosa (IMCSR), Santa Rosa, California, United States

REFERENCES:
- [Result] Church, D., & Nelms, J. (2016). Pain, range of motion, and psychological symptoms in a population with frozen shoulder: A randomized controlled dismantling study of Clinical EFT (emotional freedom techniques). Archives of Scientific Psychology, 15(1), 38-48. doi:10.1037/arc0000028
- See also: Integrative Medical Clinic of Santa Rosa — http://www.imcsr.com
- See also: Soul Medicine Institute, sponsoring organization — http://www.soulmedicineinstitute.org